CLINICAL TRIAL: NCT06089941
Title: Prospective Study of Circulating Tumor DNA Sequencing in Peripheral T-cell Lymphomas
Brief Title: Circulating Tumor DNA Sequencing in Patients With Peripheral T-cell Lymphomas
Acronym: PTCL-SEQ
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Other Study IDs: CHB23.03
Record Dates: First submitted 2023-10-09; First posted 2023-10-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T Cell Lymphoma; Next generation sequencing; circulating tumor DNA; Low-pass whole genome sequencing
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Detection of circulating tumoral DNA: Blood assessment to detect circultating tumoral DNA
  Interventions: Other: circulating tumoral DNA detection

INTERVENTIONS:
Other: circulating tumoral DNA detection — blood samples taken at diagnosis, mid-treatment, end of treatment and in the event of relapse

SUMMARY:
The purpose of this study is to assess the feasibility of analyzing circulating tumor DNA (ctDNA) as a biomarker using the shallow whole genome sequencing (lpWGS) technique coupled with deep sequencing of a targeted panel of genes (NGS), in a population of patients with newly diagnosed or relapsed/refractory peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL) are a rare and heterogeneous group of diseases resulting from the clonal proliferation of mature post-thymic lymphocytes. These T-cell neoplasms account for approximately 10-15% of all lymphomas and patients with these lymphomas have among the worst 5-year relative survivals (36%-56%, depending on prognostic factors). There are no biomarkers validated in PTCL.

Low pass whole genome sequencing (lpWGS) is an innovative molecular biology technique capable of detecting variations in the number of gene copies in patients' blood, which is a reflection of the quantity of tumor cells in the patient, lymphoma cells carrying numerous gains and deletions of certain genes at the somatic level. lpWGS is inexpensive, requires small quantities of DNA, targets the entire genome, is less time-consuming than other techniques for studying ctDNA and preliminary data in lymphomas have shown the interest of this technique. The investigators hypothesize that this study of ctDNA in PTCL will be relevant, sensitive and very informative for monitoring patients with the lpWGS technique combined with a panel of genes targeted in depth by NGS that the investigators propose to implement. This is a multicenter, prospective study, based on biological samples and clinical and imaging data to be collected.

This study will be offered to each patient suffering from PTCL, including T/NK lymphomas (NKTL) with systemic involvement (excluding cutaneous T-cell lymphomas) having an indication for systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Newly diagnosed or relapsed/refractory peripheral T-cell lymphoma (PTCL), including T/NK lymphoma (NKTL)
* Pre-therapeutic FDG PET-CT already performed
* Signed informed consent
* Patients affiliated with or beneficiaries of a health insurance plan

Exclusion Criteria:

* Cutaneous T-cell lymphomas without systemic involvement
* Pregnant or breastfeeding women
* For newly diagnosed patients: patient who has already started the first systemic treatment for their lymphoma (apart from pre-phase corticosteroid therapy which is authorized)
* For patients in a relapsed/refractory situation: Patient who has already started the new specific line of lymphoma treatment planned for the current relapsed/refractory situation (apart from pre-phase corticosteroid therapy which is authorized)
* Lack of patient consent
* Patient whose weight is less than 30 kg
* Protected adult or deprived of freedoms (under guardianship or curatorship)
* Patient unable to understand the study for any reason or to comply with the constraints of the trial (language, psychological, geographic problem, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with newly or relapse/refractory peripheral T Cell Lymphoma
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of ctDNA assessement | at the inclusion
  rate of patients considered informative (i.e. patient with at least one detectable mutation from ctDNA analysis by lpWGS and/or targeted NGS). The main objective will be achieved if the proportion of informative results is at least 90%.
Feasibility of ctDNA assessement | 8 weeks
  rate of patients considered informative (i.e. patient with at least one detectable mutation from ctDNA analysis by lpWGS and/or targeted NGS). The main objective will be achieved if the proportion of informative results is at least 90%.
Feasibility of ctDNA assessement | 16 weeks
  rate of patients considered informative (i.e. patient with at least one detectable mutation from ctDNA analysis by lpWGS and/or targeted NGS). The main objective will be achieved if the proportion of informative results is at least 90%.

SECONDARY OUTCOMES:
Concordance between ctDNA and tumor mutational profile | at the inclusion
  Description of the concordance between the mutational profile on the tumor and on plasma ctDNA at diagnosis and at relapse
Progression free survival | one year
  Time beetween inclusion and progression
Overal survival | one year
  Time beetween inclusion and death
Imaging assessment by PET-CT | 16 weeks
  Description of metabolic tumor volume before treatment, and therapeutic response (based on Lugano 2014 criteria) end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Camus, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No